CLINICAL TRIAL: NCT05773118
Title: A Unified Index to Predict the Success Probability of Myopia Control
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recent personnel changes in the research team make it unrealistic to conduct this research project.
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-597
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- orthokeratology lens (Experimental): The subjects will wear an orthokeratology lens with 3-zone reverse geometry design. The subjects are instructed to wear the lenses for at least eight hours every night and are removed during daytime hours.
  Interventions: Device: orthokeratology lens
- multifocal soft contact lens (Experimental): The subjects will wear a multifocal soft contact lens during daytime hours and remove the lens at night
  Interventions: Device: multifocal soft contact lens
- single vision spectacle (Active Comparator): The subjects will wear single vision spectacle lens as control.
  Interventions: Device: Single vision spectacles

INTERVENTIONS:
Device: orthokeratology lens — Subjects will wear orthokeratology lens at night. Axial length elongation over a period of 12-month will be recorded.
  Arms: orthokeratology lens
Device: multifocal soft contact lens — Subjects will wear multifocal soft contact lens during the day time. Axial length elongation over a period of 12-month will be recorded.
  Arms: multifocal soft contact lens
Device: Single vision spectacles — Subjects will wear single vision spectacles during the day. Axial length elongation over a period of 12-month will be recorded.
  Arms: single vision spectacle

SUMMARY:
Orthokeratology lenses (OK-lens) and multifocal contact lenses (MFCL) are optical devices designed to slow down the progression of myopia. Both treatments a long-term commitment from doctors and patients. This study aims to develop a unified index to predict the success probability of myopia control at the early stage of treatment.

DETAILED DESCRIPTION:
An Orthokeratology lens (OK-lens) is a rigid contact lens with a reverse geometry on its back surface. Overnight OK-lens wearing flattens the central cornea (creating minus power) and steepens the mid-peripheral cornea (creating plus power). During the day, this inverted pattern of peripheral corneal refraction induces relative peripheral myopic defocus on the retina to slow down the axial growth. The central portion of an MFCL is designed with minus powers to correct for distance vision, and plus power is directly added to the peripheral part of the lens. Daytime MFCL wear imposes peripheral retinal myopic defocus when the lenses are worn. An MFCL can also reduce axial growth by 52% compared to a single vision spectacle or contact lens.

Myopia control with OK-lens or MFCL requires a long-term commitment from doctors and patients to see the effect become apparent. It is paramount to estimate the probability that a patient would achieve effective control in myopic progression ideally before treatment begins or early during the course of treatment. To this end, efforts have been made to investigate the correlations between axial growth and possible contributing factors. Early research works have covered a variety of parameters at the baseline, including age, spherical equivalent (SE), corneal eccentricity, and corneal thickness. These measurements are nonspecific, indirect, and based on the assumption that their relationships to axial growth are linear, which often leads to contradictory findings and results that are hard to interpret by physicians. Therefore, in this study, we proposed a new index that takes pupil size into consideration by determining the summed relative myopic defocus dosage within the pupillary area (PMDD) to predict myopia control's success rate. This index will be determined for each eye, will be quantified one month after the lens dispensing, and will be used as the predictive variable.

ELIGIBILITY:
Inclusion Criteria:

* Older than 7 years of age or younger than 12 years of age,
* Spherical equivalent (SE) greater -1.00 D and less than-5.00 D,
* Corneal astigmatism ≤ 1.50 D,
* best-corrected visual acuity better than 20/25,
* No binocular vision dysfunction,
* No obvious angle kappa,
* No history of an OK-lens or MFCL wear or any other myopia control treatments such as atropine, application of atropine for cycloplegia during the past 30 days,
* No contact lens contraindications,
* No related ocular or systemic disease.

Exclusion Criteria:

* Younger than 7 years of age or older than 12 years of age,
* Spherical equivalent (SE) less than -1.00 D or greater than-5.00 D,
* Corneal astigmatism > 1.50 D,
* Best-corrected visual acuity less than 20/25,
* Binocular vision dysfunction,
* Obvious angle kappa,
* History of an OK-lens or MFCL wear or any other myopia control treatments such as atropine, application of atropine for cycloplegia during the past 30 days,
* Contact lens contraindications,
* Related ocular or systemic disease.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
axial length elongation | over 12 months
  The changes in axial length at the end of 12-month treatment will be computed.

SECONDARY OUTCOMES:
pupillary myopia defocus dosage | over 12 months
  The myopia defocus dosage accumulated within the pupillary area

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang D, Wen D, Zhang B, Lin W, Liu G, Du B, Lin F, Li X, Wei R. The Association between Fourier Parameters and Clinical Parameters in Myopic Children Undergoing Orthokeratology. Curr Eye Res. 2021 Nov;46(11):1637-1645. doi: 10.1080/02713683.2021.1917619. Epub 2021 Jun 6. PMID 34096430
- [Background] Xia R, Su B, Bi H, Tang J, Lin Z, Zhang B, Jiang J. Good Visual Performance Despite Reduced Optical Quality during the First Month of Orthokeratology Lens Wear. Curr Eye Res. 2020 Apr;45(4):440-449. doi: 10.1080/02713683.2019.1668950. Epub 2019 Sep 24. PMID 31526284
- [Background] Yang X, Bi H, Li L, Li S, Chen S, Zhang B, Wang Y. The Effect of Relative Corneal Refractive Power Shift Distribution on Axial Length Growth in Myopic Children Undergoing Orthokeratology Treatment. Curr Eye Res. 2021 May;46(5):657-665. doi: 10.1080/02713683.2020.1820528. Epub 2020 Sep 18. PMID 32945207
- [Background] Liu G, Wu Y, Bi H, Wang B, Gu T, Du B, Tong J, Zhang B, Wei R. Time Course of Perceived Visual Distortion and Axial Length Growth in Myopic Children Undergoing Orthokeratology. Front Neurosci. 2021 Oct 13;15:693217. doi: 10.3389/fnins.2021.693217. eCollection 2021. PMID 34720848
- [Background] Lin W, Gu T, Bi H, Du B, Zhang B, Wei R. The treatment zone decentration and corneal refractive profile changes in children undergoing orthokeratology treatment. BMC Ophthalmol. 2022 Apr 18;22(1):177. doi: 10.1186/s12886-022-02396-w. PMID 35436922
- [Background] Jiang F, Huang X, Xia H, Wang B, Lu F, Zhang B, Jiang J. The Spatial Distribution of Relative Corneal Refractive Power Shift and Axial Growth in Myopic Children: Orthokeratology Versus Multifocal Contact Lens. Front Neurosci. 2021 Jun 9;15:686932. doi: 10.3389/fnins.2021.686932. eCollection 2021. PMID 34177459
- [Background] Liu G, Jin N, Bi H, Du B, Gu T, Zhang B, Wei R. Long-Term Changes in Straylight Induced by Overnight Orthokeratology: An Objective Measure Using the Double-Pass System. Curr Eye Res. 2019 Jan;44(1):11-18. doi: 10.1080/02713683.2018.1514056. Epub 2018 Sep 10. PMID 30198800